CLINICAL TRIAL: NCT06912217
Title: Comparison of the Effects of Robotic Rehabilitation, Functional Electrical Stimulation and Occupational Therapy on Upper Extremity and Hand Functions in Tetraplegic Patients With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Hilal Buse Arslan, Principal Investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hilal Arslan 001
Record Dates: First submitted 2025-03-29; First posted 2025-04-04 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Tetraplegia/Tetraparesis
Keywords: Spinal Cord Injury; Tetraplegia; Hand Functions; Occupational Therapy; Functional Electrical Stimulation; Robotic Rehabilitation
MeSH Terms: conditions — Quadriplegia; Spinal Cord Injuries | interventions — Occupational Therapy

STUDY DESIGN:
Intervention Model Description: The study is designed as a parallel-group, open-label, prospective, randomized clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- robotic rehabilitation (Active Comparator): It is planned to provide a robotic rehabilitation program for patients in the robotic group, in addition to conventional rehabilitation for 4 weeks, with 30 minutes, 3 days a week, focusing only on their dominant upper extremities. The program will be individualized for each patient through a treatment prescription consisting of games, tailored to their joint range of motion, muscle strength, functional status, skills, and perception. The goal is for patients to perform task-specific activities on a virtual screen using an exoskeleton (Armeo Power With Manova) robotic system. The robotic systems provide three-dimensional movement ability to the extremity with motor function loss.
  Interventions: Device: Functional Electrical Stimulation; Other: occupational therapy
- Occupational therapy (Active Comparator): In the occupational therapy group, patients will receive the planned treatment in addition to conventional rehabilitation for 4 weeks, three days a week, for 30 minutes. Within the framework of this program, activities of daily living, especially self-care activities (eating, drinking, dressing, combing hair, brushing teeth, turning door handles, using remote controls, phones, and computers), as well as task-specific sensory and motor retraining and fine motor skills, will be worked on.
  Interventions: Device: robotic rehabilitation; Device: Functional Electrical Stimulation
- Functional Electrical Stimulation (Active Comparator): In the FES group, an FES bicycle program (RT300 FES leg cycle) will be applied for 4 weeks, three days a week for 30 minutes, focusing on the dominant upper extremity and hand. Electrodes will be placed on the target muscle groups. Electrodes will be placed on the elbow flexors and extensors, wrist flexors and extensors, and finger flexors and extensors. The current intensity will be adjusted according to the patient's tolerance.
  Interventions: Device: robotic rehabilitation; Other: occupational therapy

INTERVENTIONS:
Device: robotic rehabilitation — It is planned to provide a robotic rehabilitation program for patients in the robotic group, in addition to conventional rehabilitation for 4 weeks, with 30 minutes, 3 days a week, focusing only on their dominant upper extremities.
  Arms: Functional Electrical Stimulation; Occupational therapy
Device: Functional Electrical Stimulation — In the FES group, an upper extremity FES bicycle program (ADI) will be applied to the dominant upper extremity and hand, three days a week for 4 weeks.
  Arms: Occupational therapy; robotic rehabilitation
Other: occupational therapy — In the occupational therapy group, patients will receive the planned treatment in addition to conventional rehabilitation for 4 weeks, three days a week, for 30 minutes.
  Arms: Functional Electrical Stimulation; robotic rehabilitation

SUMMARY:
2. Purpose and Significance of the Study (Primary and Secondary Objectives, if any) Spinal cord injury (SCI) is a clinical condition characterized by partial or total loss of motor, sensory, and autonomic functions below the level of the lesion, depending on the severity and level of the injury, which may be caused by traumatic or non-traumatic factors.

Globally, the incidence of SCI is estimated to be 250,000-500,000 cases per year . SCI patients may be classified as tetraplegic or paraplegic according to their functional levels. In paraplegia, there is a loss of function in both lower extremities, whereas tetraplegic patients experience functional loss in all four extremities. In both groups, autonomic dysfunctions in visceral organs can also be observed depending on the severity of the injury below the lesion level.

In tetraplegic patients, loss of upper extremity and hand functions significantly reduces their level of independence in daily living activities, particularly in self-care tasks, and considerably lowers their quality of life. Therefore, upper extremity and hand rehabilitation play a crucial role in the comprehensive rehabilitation program for tetraplegic patients. Various rehabilitative modalities have been used both in clinical practice and in the literature to improve upper extremity and hand functions. The use of advanced rehabilitation technologies has increased in recent years. Studies on functional electrical stimulation (FES) for upper extremity, robotic rehabilitation, virtual reality applications, mirror therapy, and similar approaches have become more prevalent in the literature . However, there is a limited number of studies comparing the superiority of these rehabilitation techniques in tetraplegic patients, leading to insufficient data for selecting the most appropriate rehabilitative technologies in clinical practice.

This study aims to compare the effects of FES, robotic rehabilitation, and occupational therapy on upper extremity and hand functions in tetraplegic patients. Additionally, it seeks to determine which patient groups, based on their clinical and demographic characteristics, would benefit the most from each therapy and to contribute to the development of personalized rehabilitation strategies by analyzing outcomes in the acute, subacute, and chronic phases of SCI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Incomplete tetraplegia
* No cognitive impairment (Mini-Mental State Exam score ≥25)
* No significant visual deficits
* Ability to sit upright for at least 30 minutes
* No prior exposure to these treatments in the last six months

Exclusion Criteria:

* Severe upper extremity spasticity (MAS score 3-4)
* Severe shoulder pain or joint ROM restriction (>50%)
* Pre-existing neurological, rheumatological, or orthopedic conditions affecting upper extremity
* Severe cardiovascular disease
* Uncontrolled aggressive behavior
* Open wounds or infections at application sites
* Aphasia affecting comprehension
* Active deep vein thrombosis or thrombophlebitis in the upper extremity
* History of epilepsy or cyber disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Jebsen-Taylor Hand Function Test | Evaluation at Treatment Start and 4 Weeks Later
  The test consists of seven subtests:
  Writing a simple 24-letter sentence Turning over five cards Transferring small objects (e.g., buttons, jar lids, paper clips) from one container to another Simulating eating by lifting a dry bean from a plate to mouth level with a spoon Lifting empty large boxes from a table and placing them on a raised surface Lifting weighted boxes filled with objects from a table and placing them on a raised surface Stacking checkers on top of each other The patient's test completion time is recorded, and in each session, they aim to improve their previous performance.
Nine-Hole Peg Test | Evaluation at Treatment Start and 4 Weeks Later
  This test will be used to evaluate fine motor skills.
  The patient is seated at a table where the test materials are placed. The pegboard is positioned centrally on the table in front of the patient, and the pegs are placed on the side corresponding to the hand being tested.
  The patient is instructed to insert the pegs into the holes as quickly as possible, in any order, using one peg at a time, until all nine holes are filled.
  Immediately after filling all the holes, the patient is asked to remove the pegs one by one and return them to their original position without a break.
  The timer starts when the patient touches the first peg and stops when the last peg is placed. Each hand will undergo two trials, and the average time will be recorded.
Hand Grip Strength Assessment (Using a Dynamometer) | Evaluation at Treatment Start and 4 Weeks Later
  The hand grip strength of patients will be measured using a hand dynamometer.
  Measurements will be taken with the patient seated, ensuring the following positioning:
  Shoulder in adduction and close to the body
  Elbow at 90 degrees of flexion
  Wrist in 0-30 degrees of dorsiflexion and 0-15 degrees of ulnar deviation
  Thumb facing upward
  Each measurement will be repeated three times with 5-second intervals, and the average of the three measurements will be recorded in kilograms.
Pinch Grip Strength (Pinchmeter) | Evaluation at Treatment Start and 4 Weeks Later
  Measurements will be taken in a seated position with the shoulder in adduction, the elbow in 90° flexion, and the forearm in a neutral position.
  The measurements will be taken on the treated hand in three different positions: three-point, lateral, and tip-to-tip grips.
  Three-point grip strength is evaluated by applying force to the pinchmeter placed between the distal phalanx of the thumb and the pulp of the second and third fingers.
  Lateral grip strength is measured by placing the radial part of the middle phalanx of the index finger under the pinchmeter for support, while the distal phalanx of the thumb applies pressure on the pinchmeter from above.
  Tip-to-tip grip strength is measured by placing the pinchmeter between the distal tip of the thumb and the distal tip of the index finger and compressing it.
  Patients will be instructed to squeeze with maximum strength, and each measurement will be repeated three times. The averages will be recorded i
American Spinal Injury Association (ASIA): | Evaluation at Treatment Start and 4 Weeks Later
  The ASIA (American Spinal Injury Association) Spinal Cord Injury Standard Neurological Classification is a standardized system used for classifying patients with spinal cord injuries. It is an examination scale that assesses motor function, sensory function, voluntary anal contraction, and deep anal sensation.
  In the motor examination, 10 key muscle groups in both the upper and lower extremities are tested separately on the right and left sides. The sensory examination evaluates 28 dermatome areas for both light touch and pinprick sensation. A rectal examination is performed to assess voluntary anal sphincter control and the presence of deep anal sensation.
  The neurological level of injury is determined, and a distinction between complete and incomplete injury is made.

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | Evaluation at Treatment Start and 4 Weeks Later
  MAS is a six-grade scale used to assess spasticity by evaluating the resistance perceived during the passive movement of a limb. In our study, it will be used to assess spasticity in the upper extremity and hand.
ASIA Impairment Scale | Evaluation at Treatment Start and 4 Weeks Later
  Based on the results obtained from the ASIA classification system, the appropriate level for the patient is selected on the ASIA Impairment Scale, ranging from A to E.
Joint Range of Motion Assessment | Evaluation at Treatment Start and 4 Weeks Later
  The assessment will be conducted using goniometric measurements for the upper extremity and hand, following international classification standards.
Spinal Cord Injury Independence Measure (SCI Independence Measure) - Self-Care Subparameter | Evaluation at Treatment Start and 4 Weeks Later
  It is a scale used to assess functional activity limitations in spinal cord injury, evaluating a total of 17 activities, including personal care, respiration and sphincter management, and mobility. A Turkish validity and reliability study is available. In our study, the self-care subscale will be used.
  The self-care subscale consists of four parameters: eating, bathing, dressing, and grooming. The total score ranges between 0 and 20 points.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara Bilkent City Hospital, Ankara, Ankara
  - Ankara Bilkent City Hospital, Ankara, Çankaya